CLINICAL TRIAL: NCT05213832
Title: Effect of Inhalatory Sedation on Cerebral Perfusion in Subarachnoid Hemorrhage
Brief Title: Effect of Inhalatory Sedation in Subarachnoid Hemorrhage
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Maurizio Berardino, Director of Anesthesia and Intensive Care Unit Departement, A.O.U. Città della Salute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0076379
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Subarachnoid Hemorrhage; Aneurysmal Subarachnoid Hemorrhage
Keywords: perfusion; isofluorane; inhalatory; sedation
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhalatory group (Experimental): Patience with severe SAH (WFNS > 3) are enrolled in the study. In these patients we administered a inhalatory dose of Isofluorane
  Interventions: Drug: Isoflurane Inhal Soln

INTERVENTIONS:
Drug: Isoflurane Inhal Soln — Administration of isofluorane in patients with severe SAH

SUMMARY:
The aim of this study is to evaluate the effect of inhalational sedation on cerebral perfusion in patients with SAH.

It will evaluate whether the administration of isofluorane, by inducing direct vasodilation in the cerebral parenchyma, can improve the cerebral perfusion rates.

Perfusional CT will be used to study the variation of cerebral blood flow to rule out the vasodilatory effect on territories with different cerebrovascular reactivity aggravating the phenomena of distrectual hypoperfusion (theft theory).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of non-traumatic SAH
* Neurological and/or systemic presentation that requires support of vital functions and sedation. This occurs for a WFNS score (World Federation of Neurosurgical Societies) ≥ 3.
* Possibility of ICP monitoring through EVD which is necessary in case of acute hydrocephalous. In case of the neurosurgeon do not indicate the positioning of the EVD, an intraparenchymal catheter will be positioned for the ICP monitoring.
* Patients with vasospasm (area of cerebral blood flow under 30% of the best value detected in the brain of the patients at the first CT scan). This exam will be performed at 2° - 3° day post event.
* Acceptance of informed consent.

Exclusion Criteria:

* Documented outcomes of cerebrovascular disease
* Patients with acute heart failure related to ESA
* State of pregnancy
* Patients with CLCR < 30 mL/min

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow recondtion | 20 minutes
  The percentage of subjects who had a flow recondition at the second CT at least 50% of the best value detected in the first perfusion CT scan

SECONDARY OUTCOMES:
Changes in intracranial pressure during isoflurane delivery | 20 minutes
  We evaluate if isofluorane create an increase in ICP trough continuous monitoring.
Changes in blood pressure during isoflurane delivery | 20 minutes
  By its vasodilatatore effect, we monitored punctually if mean arterial blood pressure will increase during isofluorane delivery

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Berardino, MD, Principal Investigator — AOU Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza - Presidio CTO, Torino, Italy